CLINICAL TRIAL: NCT06440083
Title: Pre-warning Risk Scoring System for Sudden Cardiac Death
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jingfeng Wang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2023-177-01
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Sudden Cardiac Death
Keywords: Sudden Cardiac Death; Cohort study
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to identify potential indicators for pre-warning of sudden cardiac death (SCD), including clinical biochemistry markers, electrocardiogram, echocardiography, MRI and CT imaging values, genetic markers and so on, and further construct a series of multi-parameter assessments of SCD early screening.

DETAILED DESCRIPTION:
In the past few decades, evidence-based drug and surgical treatment strategies have significantly improved the prevention of sudden cardiac death (SCD), however, a large number of patients with cardiovascular disease still face high risk of SCD, the prognosis of these high-risk SCD patients are still uncertain. Therefore, clinical physicians might need to move towards a multi-parameter assessment of SCD risk pre-warning. Several parameters for risk stratification of arrhythmia, including clinical biochemistry markers, electrocardiogram, echocardiography, imaging, and genetic markers, are crucial for accurate assessment of SCD risk stratification. In addition, the integration of cardiac magnetic resonance parameters and specific CT and ECG information is a future research trend for implementing risk stratification of malignant arrhythmias. In order to further explore the possibility of early warning of SCD, this study aims to include subjects with potential SCD risks, collect relevant potential SCD warning indicators, and then construct an SCD prewarning score system. Afterwards, the investigators will continuously improve the SCD warning score system based on follow-up information, and ultimately summarize an effective set of SCD warning scores and apply them to clinical practice, striving to achieve early warning of SCD and benefiting more people at risk of SCD.

ELIGIBILITY:
Inclusion Criteria:

The subjects with the following diagnosis of one or more cardiovascular diseases:

1. Coronary heart disease If there is a history of coronary heart disease or a new diagnosis of coronary heart disease, or with a report of coronary angiography that indicates at least one vascular stenosis>50%. Diagnosis includes chronic coronary syndrome (stable angina, ischemic cardiomyopathy, and occult coronary heart disease) and acute coronary syndrome (unstable angina, ST-segment elevation myocardial infarction and non-ST-segment elevation myocardial infarction).
2. Heart failure Individuals with a history of heart failure or newly diagnosed heart failure, including heart failure with reduced ejection fraction (HFrEF, left ventricular ejection fraction (LVEF) ≤40%)、intermediate heart failure (HFmrEF, LVEF 41%-49%，with evidence of spontaneous or excitable increase in left ventricular filling pressure), and ejection fraction preserving heart failure (HFpEF, LVEF≥50%, there is evidence of spontaneous or excitable increase in left ventricular filling pressure).
3. Genetically related cardiomyopathy or arrhythmia Cardiomyopathy includes hypertrophic cardiomyopathy (DCM), dilated cardiomyopathy (HCM), arrhythmogenic right ventricular cardiomyopathy (ARVC), inflammatory cardiomyopathy (myocarditis, sarcoidosis, Chagas disease). Hereditary arrhythmias include long QT syndrome, short QT syndrome, Brugada syndrome, idiopathic ventricular fibrillation, catecholamine sensitive polymorphic ventricular tachycardia (CPVT), early repolarization syndrome, etc.

2) Sign an informed consent form.

Exclusion Criteria:

1. Age<16 years old;
2. Refusal to the follow-up visits;
3. Individuals with severe mental disorders who are unable to express their wishes;
4. Other obvious physical diseases and abnormal laboratory test results;
5. Patients deemed unsuitable for participation in this study by the supervising physician.

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with potential high-risk of sudden cardiac death.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sudden cardiac death | Baseline and to the 1-year, 2-year, 5-year follow-up
  Identify participants who die by cardiovascular diseases during follow-up period

SECONDARY OUTCOMES:
All-causes death | Baseline and to the 1-year, 2-year, 5-year follow-up
  Identify participants who die during follow-up period
Recurrence of cardiovascular disease | Baseline and to the 1-year, 2-year, 5-year follow-up
  Identify participants who with recurrence of cardiovascular disease during follow-up period
Cardiac arrest | Baseline and to the 1-year, 2-year, 5-year follow-up
  Identify participants who suffer sudden cardiac arrest during follow-up period
Major cardiovascular events | Baseline and to the 1-year, 2-year, 5-year follow-up
  Identify participants who suffer incident major cardiovascular events during follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Jingfeng Wang, M.D.,Ph.D., Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guanzhou, Guangdong, China